CLINICAL TRIAL: NCT03847077
Title: Randomized Trial of a Patient Education Tool For Leiomyoma
Brief Title: Trial of a Patient Education Tool For Leiomyoma
Acronym: PETAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Linda Yang, MD, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207033
Record Dates: First submitted 2019-02-08; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Uterine Leiomyoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPad counseling (Experimental): Women with leiomyomata confirmed on imaging who presented as a new patient to the gynecology clinic at a single institution were randomized to receive multimedia counseling using the drawMD OB/GYN iPad application
  Interventions: Behavioral: iPad counseling
- Standard counseling (Active Comparator): Women with leiomyomata confirmed on imaging who presented as a new patient to the gynecology clinic at a single institution were randomized to receive standard counseling.
  Interventions: Behavioral: Standard Counseling

INTERVENTIONS:
Behavioral: iPad counseling — Women with leiomyomata confirmed on imaging who presented as a new patient to the gynecology clinic at a single institution were randomized to receive multimedia counseling using the drawMD OB/GYN iPad application.
  Arms: iPad counseling
Behavioral: Standard Counseling — Women with leiomyomata confirmed on imaging who presented as a new patient to the gynecology clinic at a single institution were randomized to receive standard counseling.
  Arms: Standard counseling

SUMMARY:
The goal of this study was to assess whether using a multimedia tool would enhance patient education and counseling on uterine leiomyomata.

DETAILED DESCRIPTION:
Women with leiomyomata confirmed on imaging who presented as a new patient to the gynecology clinic at a single institution were randomized to receive either standard counseling or multimedia counseling using the drawMD OB/GYN iPad application. Participants completed a pre-counseling questionnaire, received the designated method of counseling, and then completed a post-counseling questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant
* English speaking
* Women aged 18-60 years
* presence of fibroids confirmed on imaging
* no confirmed or suspicion of malignancy

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Change in patient knowledge scores | Day 1
  Patients were asked baseline knowledge questions about fibroids prior to receiving physician counseling. Patients were randomized to iPad counseling or standard counseling groups. After the counseling session, patients answered similar knowledge questions about fibroids. The pre-counseling and post-counseling scores will be compared for each group. Generalized estimating equations were used to test whether any change in knowledge from pre-counseling to post-counseling was dependent on the participant's intervention assignment.
Patient satisfaction post-counseling | Day 1
  Patients completed a Likert scale questionnaire (1 = Very Dissatisfied, 2 = Dissatisfied, 3 = Neutral, 4 = Satisfied, 5 = Extremely Satisfied) to evaluate satisfaction with assigned counseling method.
Patient anxiety pre-couseling | Day 1
  Participants completed a Likert scale questionnaire (1 = Not at all, 2 = Somewhat, 3 = Moderately, 4 = Very Much) about their anxiety related to fibroids prior to receiving physician counseling.
Patient anxiety post-couseling | Day 1
  Participants completed a Likert scale questionnaire (1 = Not at all, 2 = Somewhat, 3 = Moderately, 4 = Very Much) about their anxiety related to fibroids after receiving physician counseling.